CLINICAL TRIAL: NCT07021404
Title: The Epidemiology of Suicide Attempts and Suicidal Thoughts in Flanders
Acronym: BC-03869
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-03869
Record Dates: First submitted 2025-03-17; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Suicidal Ideation; Suicide Attempt; Multicenter Study; Epidemiological Study; Suicidal Behavior
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted | interventions — Guidelines as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Individuals who presented with suïcidale behavior to Hospitals and other healthcare institutions
  Interventions: Other: Semi-structured interview (Guideline for Suicide care and Evaluation =LOES)

INTERVENTIONS:
Other: Semi-structured interview (Guideline for Suicide care and Evaluation =LOES) — A semi-structured interview is utilized in general hospitals and other healthcare institutions by clinicians and nurses as part of the psychosocial assessment, with the aim of collecting standardized data on episodes of self-harm and individuals experiencing suicidal ideation.
  The interview consists of two parts:
  Part 1 is administered shortly after admission to the healthcare facility due to an episode of self-harm or reported suicidal thoughts. It is conducted by a trained nurse or psychologist. This section collects demographic information, characteristics of the self-harm episode, history of self-harm behavior, perceived social support, level of hopelessness, and current suicidal ideation.
  Part 2 focuses on a more in-depth exploration of the individual's psychological state. It assesses underlying motives for the self-harm or suicidal thoughts, perceived personal and interpersonal problems, and current and current thoughts of self-harm.

SUMMARY:
The objective of this study is to collect data in Flanders on the incidence of suicide attempts and suicidal ideation across various healthcare settings. The study also aims to assess the proportion of individuals who receive adequate aftercare following a suicide attempt and to systematically document the methods and means used in suicidal behavior.

DETAILED DESCRIPTION:
This study involves the registration of the frequency and characteristics of suicidal thoughts and suicide attempts among individuals presenting to healthcare services (including general hospitals, psychiatric hospitals, mobile crisis teams, and general practitioners). Participants will be evaluated using a semi-structured interview: the Guideline for Suicide Care and Evaluation (LOES).

The primary objective is to collect detailed data on individuals with suicidal behavior-including suicidal ideation and suicide attempts-using the LOES instrument. This approach allows for the collection of comprehensive information about suicidal individuals in Flanders and the suicidal processes affecting them.

The LOES comprises two components:

1. Basic Assessment The initial assessment occurs shortly after the individual presents at a healthcare institution. During this interview, an emergency nurse, physician, psychologist, or psychiatrist evaluates the individual's cognitive functioning, judgment, emotional state, observable behavior, potential mental health disorders, history of self-harm or suicidal behavior, social support, level of hopelessness, and willingness to engage in follow-up care. Sociodemographic data and details about the current and any previous suicide attempts are also recorded.

   The goals of this assessment are:
   * To ensure the individual feels heard and taken seriously.
   * To determine the appropriate timing for a more comprehensive risk assessment based on the initial findings.
2. Further Exploration of Suicidality This second phase is conducted by a nurse, psychologist, or psychiatrist. It includes a more in-depth evaluation of the individual's risk factors and treatment needs. Standardized questions cover topics such as suicidal intent, suicidal ideation and concrete planning, motivations for self-harm or suicidal thoughts, ambivalence, experienced life problems, psychiatric history, potential substance use, coping strategies, and care needs of both the individual and their immediate environment.

Based on the data collected through the LOES, a structured and well-supported risk formulation can be established.

ELIGIBILITY:
Inclusion Criteria:

* Everyone who is admitted alive to the emergency department after a suicide attempt is included. All methods used during the suicide attempt are included. Regarding the method of suicide attempts, a distinction is made between self-injury (hanging, strangulation, drowning, stab and cut wounds, jumping from a height, etc.) and self-poisoning (ingestion of (psycho)pharmaceuticals, drugs, alcohol, chemicals, or other harmful substances).
* Everyone who is admitted with suicidal thoughts

Exclusion Criteria:

* Accidental overdose, e.g., someone taking medication for a medical condition without any intent to harm themselves
* Alcohol intoxication without any intent to harm oneself
* Accidental overdose involving party drugs
* Individuals who were deceased upon arrival at the hospital due to suicide

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of individuals who are admitted to hospitals or other healthcare institutions, clinic of University Hospital Ghent, A-zorg Aalst, Vitaz Sint-Niklaas, AZ Herentals, AZ Oudenaarde, AZ Sint-Lucas Gent, AZ Sint Vincentius Deinze, AZ Sint Blasius Dendermonde, AZ Jan Palfijn Gent, AZ Alma Eeklo, AZ Groeninge Kortrijk, AZ Oostende, OLV v Lourdes Waregem, AZ Sint Jan Brugge, AZ West Veurne, AZ Sint Lucas Brugge, Jan Yperman ziekenhuis, Sint Andriesziekenhuis Tielt, Sint-Jozefskliniek Izegem, AZ Delta Roeselare, AZ Sint Maria Halle, AZ diest, AZ Klina Brasschaat, AZ Monica Deurne, AZ Sint Maarten Mechelen, AZ Voorkempen Malle, Ziekenhuis Geel, Heilig Hart Lier, Universitair Ziekenhuis Antwerpen, Imeldaziekenhuis Bonheiden, ZSA-UKJA Antwerpen, Sint-Trudo Sint-Truiden, ZOL Genk, Psychiatrisch ziekenhuis Bilzen-Hoeselt.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2006-12-31 (Actual); Primary Completion 2033-03-31 (Estimated); Study Completion 2033-03-31 (Estimated)

PRIMARY OUTCOMES:
Baseline Demographic and Socioeconomic Characteristics | Day 1
  Sociodemographic information will be collected via standardized intake forms during the initial assessment interview. The following variables will be recorded:
  * Date of birth (continuous, in DD/MM/YYYY format)
  * Gender (Male / Female / X)
  * Marital status (Unmarried / Officially cohabitating / Married / Divorced / Widowed)
  * Housing situation (Alone / Not alone)
  * Presence of children (Yes / No)
  * Economic activity status (Economically active / Unemployed / Economically inactive)
    * If economically inactive: Pupil or student / Disability due to physical or psychological problems / Retirement / Other (specify) Profession (open text, if applicable)
  * School situation (if student):
    * Primary education
    * Secondary education (ASO / TSO / BSO / KSO / BuSO)
    * Higher education or university
    * Other (specify) All responses will be recorded and coded for analysis. Categorical variables will be summarized using frequency and percentage. Open-ended responses will be described narratively
Baseline Demographic, Socioeconomic and Clinical Admission Characteristics | Day 1
  Additional personal and contextual characteristics will be collected during the initial assessment interview. These include:
  Pregnancy status (Yes / No)
  Country of birth of the participant, their mother, and their father (Belgium / Other - specify)
  Current medication: Open-ended question regarding all prescribed or self-used medications at time of intake.
  Reason for admission (Suicidal thoughts / Suicide attempt)
  All categorical variables will be recorded using predefined categories. Open-text fields (e.g., country of birth, medication list) will be thematically categorized post-hoc where applicable. These variables are used to describe the population and examine their relationship with clinical outcomes.
Method of Suicide Attempt Classified by ICD-10 Category | Day 1
  The method of suicide attempt will be assessed through a semi-structured interview and classified according to the relevant ICD-10 codes for intentional self-harm (e.g., X60-X84). Each participant's attempt will be categorized based on the specific method used (e.g., poisoning, cutting, jumping, hanging), as defined by ICD-10 classification.
Assessment of Current Emotional State (Open-Ended Response) | Day 1
  Participants will be asked the open-ended question:
  "How are you feeling right now?" Responses will be collected verbatim during a clinical interview. A qualitative content or thematic analysis will be performed to identify and categorize emotional states (e.g., anxious, sad, calm, angry). The number and percentage of participants reporting each emotional category will be reported.
Suicidal Ideation Attributes (Modified SIDAS) | Day 1
  A modified version of the Suicidal Ideation Attributes Scale (SIDAS) will be used to assess the presence and characteristics of suicidal ideation in the past month. The following six items will be included:
  * Current suicidal thoughts: Response: Yes / No.
  * Frequency of suicidal thoughts in the past month
  * Duration of suicidal thoughts
  * Perceived control over suicidal thoughts
  * Emotional suffering due to suicidal thoughts
  * Functional interference (e.g. with work or household tasks)
  * Proximity to a suicide attempt in the past month (only asked if ideation present, not in case of actual attempt).
  This version retains the conceptual dimensions of the original SIDAS but uses predefined categorical response scales instead of numerical ratings. Results will be analyzed using frequency distributions and, where appropriate, ordinal scales. This adapted version allows for structured yet clinically nuanced evaluation of suicidal ideation during intake.
Assessment of Suicidal Planning and Intent (Mixed-Methods Interview) | Day 1
  Suicidal planning and intent will be assessed through a structured set of questions combining categorical responses and open-ended fields. The following domains will be evaluated:
  Presence of a current suicide plan (categorized as: no thoughts, thoughts without plan, detailed plan)
  Method(s) considered (open-ended response)
  Availability of method (Yes/No)
  Degree of preparation (No preparation, Minimal preparation, Extensive preparation)
  Timing and delay of planned action (open-ended response)
  Categorical data will be analyzed descriptively (counts and percentages per category). Open-ended responses will undergo thematic analysis to identify patterns in methods considered and perceived urgency or control over suicidal intent.
History of Suicidal Behavior and Post-Attempt Treatment (Structured Interview) | Day 1
  Participants will be asked a structured set of questions to assess the history of suicidal behavior and care received following previous suicide attempts. The following aspects will be recorded:
  Number of lifetime suicide attempts (0, 1, 2, 3, ≥4)
  Time since last attempt (≤6 months, 6-12 months, >12 months)
  Psychological treatment received after attempt (Yes/No)
  Satisfaction with treatment (Yes/No)
  Type of provider or setting (e.g., psychiatrist, school guidance center, residential care, mental health center, other)
  Whether the attempt required medical treatment (Yes/No) and location (e.g., hospital, general practitioner, other)
  Method used in previous attempt(s) (open-ended)
  Categorical data will be summarized using frequencies and percentages. Open-ended responses on method used will be analyzed qualitatively and grouped by ICD-10 method category (e.g., poisoning, cutting, jumping).
History and Recency of Self-Harming Behavior (Structured Interview) | Day 1
  Participants will be asked whether they have ever deliberately hurt or injured themselves (Yes/No). If the response is Yes, they will be asked to indicate when they last engaged in self-harming behavior:
  < 6 months ago > 6 months ago
  Responses will be recorded categorically to assess lifetime presence and recency of non-suicidal self-injury (NSSI) or deliberate self-harm.
Perceived Social Support and Help-Seeking Behavior (Semi-Structured Interview) | Day 1
  Social support will be assessed using a semi-structured interview consisting of both categorical and open-ended questions, focusing on:
  Perceived emotional support: "Do you feel there are people who care about you?" (Yes/No)
  Identified source(s) of support: Open-ended response if Yes
  Availability of support when struggling: (Not inclined to seek support / No / Yes)
  Identified support figure: Open-ended response if Yes
  Actual help-seeking behavior: (No / Sometimes / Yes)
  Open-ended responses (e.g., to whom the participant turns) will be categorized using inductive thematic coding. Categorical responses will be summarized as frequencies and proportions.
Participant's Experience of Hopelessness (Open-Ended Response) | Day 1
  Participants will be asked the following open-ended questions:
  "Do you feel completely stuck, as if there is no way out?" "Do you feel hopeless, like there's no way out of your situation?" "Is there anything that might help you get through this period?" Responses will be collected in written form. Qualitative analysis (e.g., thematic analysis or content coding) will be used to identify recurring expressions of hopelessness or related emotional states. Results will be reported as the number and percentage of participants expressing each identified theme.
Openness to Professional Help When Experiencing Suicidal Thoughts | Day 1
  Participants will be asked about their willingness to engage in professional help when struggling with suicidal thoughts. The question is phrased as:
  "When struggling with suicidal thoughts, it is recommended to get professional help. Would you be open to have a conversation with [healthcare provider] to gain more insight into the things you are struggling with and possible next steps?"
  Response options are:
  * Does not want professional help
  * Neutral
  * Is open to professional help
  Responses will be recorded categorically and reported as frequencies and proportions across the three levels.
Suicide Intent Severity Assessed by Suicide Intent Scale (SIS) | Day 1
  The severity of intent during the most recent suicide attempt will be assessed using the Suicide Intent Scale (SIS). The SIS is a 8-item clinician-administered scale evaluating objective circumstances and subjective expectations associated with the attempt.
  Each item is scored from 0 to 2 (range total score: 0-16), with higher scores indicating greater suicidal intent.
  Scores will be reported as continuous outcomes (mean, SD), and optionally categorized (e.g., low intent: ≤5; high: >6).
Motives for Suicide Attempt Based on Structured Clinician Classification | Day 1
  Motives for the suicidal behavior will first be explored through an open-ended question:
  "What motives did you have for your suicide attempt / suicidal thoughts?"
  Based on the participant's narrative, the clinician will categorize the motives using a predefined set of thematic categories:
  * Internal conflict (e.g., emotional overwhelm, self-punishment, feeling of failure)
  * Interpersonal motives (e.g., desire to be heard, influence others, show love, revenge)
  * Death wish
  * Magical thinking (e.g., rebirth, reunion with deceased)
  Multiple categories may be selected per participant. Open-text responses will be retained for qualitative analysis; category selections will be summarized as frequencies and proportions.
Sources of Ambivalence Toward Suicide Attempt (Open-Ended Interview Question) | Day 1
  Participants will be asked the open-ended question:
  "What is currently stopping you from attempting suicide?"
  Responses will be documented verbatim. No predefined answer categories will be provided. The data will be used for qualitative analysis of protective factors, barriers, or ambivalent thoughts associated with suicidal ideation or behavior.
Presence and Duration of Stressful or Traumatic Life Events (Clinician-Coded Intake Observation) | Day 1
  During the assessment, clinicians will code the presence and estimated duration of any significant life events or psychosocial stressors spontaneously reported by the participant, based on a predefined list of known suicide-related risk factors. These include:
  * Health-related: psychiatric symptoms, physical illness, disability
  * Loss-related: death or illness of a significant person, suicide or suicide attempt of a significant other
  * Trauma: abuse (physical/emotional/sexual), neglect, assault
  * Social/relational: problems with parents, children, partner, friends, bullying
  * Environmental stressors: financial, housing, work/school, legal, identity-related problems
  Each event is coded by the clinician if mentioned, and the duration of suffering related to each event is estimated using a 3-point scale:
  1. = weeks
  2. = months
  3. = years
Substance Use Risk Assessed by CRAFFT Screening Tool | Day 1
  Substance use risk will be assessed using the CRAFFT Screening Interview, a validated 6-item questionnaire designed to identify risky substance use behaviors among adolescents and young adults. Each item is scored 0 (No) or 1 (Yes), resulting in a total score ranging from 0 to 6. A score of ≥2 indicates high risk of problematic substance use.
History of Mental Health Problems and Prior Treatment (Categorical and Narrative Assessment) | Day 1
  Participants will be asked whether they have experienced previous mental health problems and whether they sought or received professional treatment. Responses will be recorded using the following categories:
  * No previous mental health problems
  * Yes, previous mental health problems but no treatment
  * Yes, previous mental health problems and received treatment
  For those indicating previous problems, clinicians will document:
  Nature of past mental health issues (open-ended) Type of treatment received (e.g., psychologist, psychiatrist, residential care) and experience with care (open-ended) Whether a formal psychiatric diagnosis was given (open-ended)
  Open text responses will be used for qualitative description and may be thematically coded if relevant to the analysis.
Coping Strategies in Response to Stress (Narrative and Structured Clinician Assessment) | Day 1
  Participants will be asked an open-ended question exploring how they typically deal with stress and difficult emotions:
  "How do you deal with problems in general? What do you do when you are worried or upset? What helps you keep going?"
  The clinician will document the participant's narrative response and will also indicate the presence or absence of specific coping behaviors based on a predefined checklist:
  * Talks to someone about it
  * Blames self for being in trouble
  * Gets angry
  * Withdraws/stays in room
  * Reflects on previous coping experiences
  * Uses alcohol or drugs
  * Avoids thinking about worries
  * Tries to sort things out Multiple behaviors can be selected per participant.
Perceived Positive and Negative Future Events (Open-Ended Interview Questions) | Day 1
  Participants will be asked two open-ended questions to explore their short-term future outlook:
  "Are there any positive things or events in the near future that could affect your suicidal thoughts?"
  "Are there any negative things or events in the near future that could affect your suicidal thoughts?"
  Responses will be documented verbatim. No predefined response categories are used. Responses will provide insight into the participant's subjective experience of hope, anticipatory stress, or protective/risk factors linked to future-oriented thinking.
Patient-Reported Care Needs and Expectations (Open-Ended Interview Response) | Day 1
  Participants will be asked open-ended questions regarding their perceived care needs and expectations for support.
  Formal Care Setting: The participant's responses will be categorized into care delivery modes such as ambulatory care, residential care, general practitioner (GP) involvement.
  Content of Care: The narrative responses will be analyzed for themes related to the nature of care needed, including but not limited to psychological support (individual or group therapy), practical assistance, need for rest or stabilization.
  Responses will be documented verbatim and later coded using thematic analysis.
Post-Assessment Care Pathways and Treatment Agreements | Day 1
  Following the clinical intake, the treating clinician will document the planned care pathway for the participant by selecting one or more of the following options:
  No further treatment
  * Discharge (advised) (e.g., returning home)
  * Discharge (counter-advised) (e.g., patient runs away)
  * Return to another facility (e.g., detention unit, sheltered housing, medical pedagogical institution)
  Outpatient treatment (e.g., psychotherapy)
  Inpatient treatment
  * Somatic unit
  * Emergency psychiatry
  * Child/adolescent psychiatric crisis unit
  * Child/adolescent psychiatric unit
  * Psychiatric Ward General Hospital (PAAZ)
  * Psychiatric Hospital (PZ) / Psychiatric Care Home (PVT)
  * Other settings (specify): ____________________________
  In addition, any concrete treatment agreements made with the participant will be documented in free text. Monitoring these aspects is essential for evaluating care continuity, adherence to treatment plans, and subsequent clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Portzky, Prof, Principal Investigator — University Ghent
Locations (33):
- Belgium (33):
  - Azorg, Aalst
  - Ziekenhuis aan de Stroom (UKJA), Antwerp
  - Universitair ziekenhuis Antwerpen, Antwerp
  - Psychiatrisch ziekenhuis Bilzen-Hoeselt, Bilzen
  - Imeldaziekenhuis, Bonheiden
  - AZ Klina, Brasschaat
  - AZ sint Jan, Bruges
  - AZ sint Lucas, Bruges
  - AZ Sint Vincentius, Deinze
  - AZ Sint Blasius, Dendermonde
  - AZ Monica, Deurne
  - AZ Diest, Diest
  - AZ Alma, Eeklo
  - Ziekenhuis Geel, Geel
  - Ziekenhuis Oost Limburg, Genk
  - AZ Jan Palfijn, Ghent
  - AZ Sint-Lucas, Ghent
  - AZ Sint Maria, Halle
  - AZ Herentals, Herentals
  - Jan Yperman ziekenhuis, Ieper
  - Sint-Jozefskliniek, Izegem
  - AZ Groeninge, Kortrijk
  - Heilig Hart Lier, Lier
  - AZ Voorkempen, Malle
  - AZ Sint Maarten, Mechelen
  - AZ oostende, Ostend
  - AZ Oudenaarde, Oudenaarde
  - AZ Delta, Roeselare
  - VITAZ, Sint-Niklaas
  - Sint-Trudo ziekenhuis, Sint-Truiden
  - Sint Andriesziekenhuis, Tielt
  - AZ West, Veurne
  - O.L.V. van Lourdes ziekenhuis Waregem, Waregem

IPD SHARING:
Plan to Share IPD: No
The investigators have decided not to share the IDP collected throughout the trial due to concerns over participant privacy and data confidentiality. Despite efforts to anonymize the data, there remains a risk that sensitive personal information could be inadvertently disclosed.

REFERENCES:
- [Background] Vancayseele N, Portzky G, van Heeringen K. Increase in Self-Injury as a Method of Self-Harm in Ghent, Belgium: 1987-2013. PLoS One. 2016 Jun 1;11(6):e0156711. doi: 10.1371/journal.pone.0156711. eCollection 2016. PMID 27249421
- [Background] de Beurs D, Vancayseele N, van Borkulo C, Portzky G, van Heeringen K. The association between motives, perceived problems and current thoughts of self-harm following an episode of self-harm. A network analysis. J Affect Disord. 2018 Nov;240:262-270. doi: 10.1016/j.jad.2018.07.047. Epub 2018 Jul 27. PMID 30086470
- [Background] Vancayseele N, Rotsaert I, Portzky G, van Heeringen K. Medication used in intentional drug overdose in Flanders 2008-2013. PLoS One. 2019 May 2;14(5):e0216317. doi: 10.1371/journal.pone.0216317. eCollection 2019. PMID 31048918
- See also: The page refers to the semi-structured interview and more information about the study — http://www.zelfmoord1813.be